CLINICAL TRIAL: NCT07353944
Title: Assessment of Patient Satisfaction With Transcutaneous Tibial Nerve Stimulation in a County Hospital System
Brief Title: TTNS vs PTNS in a County Hospital System.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Tajnoos Yazdany, M.D., Principal Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-32833-01
Record Dates: First submitted 2026-01-16; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2019-03

CONDITIONS: Overactive Bladder
Keywords: overactive bladder; OAB; PTNS; percutaneous tibial nerve stimulation; TTNS; transcutaneous tibial nerve stimulation; county hospital; underserved
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Investigator, Outcomes Assessor
Masking Description: After randomization, patients and care providers will not be blinded, however investigators will be blinded to the results of the survey instruments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Percutaneous tibial nerve stimulation (PTNS) (Active Comparator): Participants undergo weekly 30-minute percutaneous tibial nerve stimulation in our clinic. The PTNS device is a neuromodulation system comprised of an external signal generator attached to one electrode that is placed on the patient's foot, and the other to an acupuncture needle that is inserted in the patient's inner ankle. It delivers a low electrical signal (20 Hz, 200ms pulse width) to the posterior tibial nerve, adjusted to the participant's perception of stimulation without pain.
  Interventions: Device: Tibial nerve stimulation
- Transcutaneous tibial nerve stimulation (TTNS) (Experimental): Participants receive a TENS unit and are taught how to conduct TTNS therapy at home at their recruitment visit. The TENS unit is a neuromodulation system comprised of an external signal generator attached to one electrode that is placed on the patient's foot, and the other to an electrode patch that is inserted in the patient's inner ankle. It delivers a low electrical signal (20 Hz, 200ms pulse width) to the posterior tibial nerve, adjusted to the participant's perception of stimulation without pain. They will be instructed to conduct this therapy every other day at home.
  Interventions: Device: Tibial nerve stimulation

INTERVENTIONS:
Device: Tibial nerve stimulation — neuromodulation therapy for overactive bladder that targets the posterior tibial nerve
  Other Names: PTNS; TTNS

SUMMARY:
The goal of this clinical trial is to study whether transcutaneous tibial nerve stimulation (TTNS) is a feasible and satisfactory treatment for overactive bladder in Urogynecology patients who receive their care at a county hospital.

Researchers will compare outcomes with TTNS to patients who undergo percutaneous tibial nerve stimulation (PTNS).

The main questions it aims to answer are:

* Is TTNS non-inferior to PTNS in terms of OAB symptom severity?
* Are patients as satisfied with TTNS as they are with PTNS?
* Are patients' symptoms improved with TTNS?

Participants will:

* either undergo PTNS or be taught how to do TTNS therapy at home
* complete surveys about their bladder symptoms and satisfaction with treatment

DETAILED DESCRIPTION:
Patients who consent to this study will be randomly assigned to either receive PTNS in clinic weekly, or TTNS every other day at home. The severity of their overactive bladder symptoms and satisfaction with treatment will be assessed before starting treatment as well as 6 weeks, 12 weeks and 6 months after starting treatment. The results of these surveys will be compared between groups to determine whether TTNS is non-inferior to PTNS in this particular patient population.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 - 90 years old
* patient of the Urogynecology clinic at Harbor UCLA medical center
* diagnosis of overactive bladder
* patient elects non-pharmacologic treatment of overactive bladder
* English or Spanish speaking
* able to consent and participate in research

Exclusion Criteria:

* cognitive impairment or diagnosis of dementia
* diagnosis of neurogenic bladder
* prior midurethral sling procedure
* use of an electronic pacemaker
* current pregnancy
* incarcerated persons

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2017-01-18 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
ICIQ-OAB score | Baseline, 6 weeks, 12 weeks, 6 months post treatment initiation
  OAB symptom severity

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks, 12 weeks, 6 months post treatment initiation
  Patient satisfaction with the intervention (Y/N; would you recommend it to others?)
PGI-I | 6 weeks, 12 weeks, 6 months post treatment initiation
  Patient global assessment of overall improvement, graded on a scale of 1-7
Compliance | 6 months post treatment initiation
  Number and percentage of PTNS visits (PTNS arm); Patient reported number of self-administered TTNS treatments per week

CONTACTS AND LOCATIONS:
Locations (1):
- Harbor UCLA Medical Center, Torrance, California, United States